CLINICAL TRIAL: NCT07197775
Title: Endogenex PULSE Registry
Brief Title: Post-market SUrveiLlance RegiStry for the Endogenex System (Endogenex PULSE Registry)
Status: Not yet recruiting | Type: Observational
Sponsor: Endogenex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1419
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Type2Diabetes; Diabetes Mellitus, Type 2; Type 2 Diabetes; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Endogenex System Treated: Participants treated with the Endogenex System

SUMMARY:
This registry is designed to collect long-term data and support ongoing post-market surveillance of real-world data for the Endogenex System.

DETAILED DESCRIPTION:
This is an observational registry that is designed to facilitate long-term patient follow-up for up to 5 years after an Endogenex procedure. It is structured to enable systematic longitudinal data collection on the safety and long-term clinical outcomes associated with the Endogenex System.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Have been treated with the Endogenex System
* Consented to participate in the Endogenex PULSE Registry

Exclusion Criteria:

* Unwilling or unable to attend study visits
* Unwilling or unable to provide medical records to study sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been treated with the Endogenex System.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2032-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 5 years
  Incidence of device-related and/or procedure-related adverse events

IPD SHARING:
Plan to Share IPD: No